CLINICAL TRIAL: NCT00042666
Title: A Phase 2 Evaluation of Oral LY317615 in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Oral LY317615 in Relapsed or Refractory Diffuse Large B-Cell Lymphomas.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4849; H6Q-MC-JCAI (Other: Eli Lilly and Company); NCT00054080 (obsolete NCT alias)
Record Dates: First submitted 2002-08-02; First posted 2002-08-06 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY317615 (Experimental): 500 milligrams (mg), oral, daily (QD), up to six (6) 28-day cycles
  Interventions: Drug: LY317615

INTERVENTIONS:
Drug: LY317615 — 500 mg, oral, QD, up to six 28 day cycles
  Other Names: enzastaurin

SUMMARY:
This study will measure the effectiveness and any side effects of LY317615 in participants with diffuse large B-cell lymphoma (DLBCL: a sub-type of Non-Hodgkins Lymphoma).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of recurrent or refractory DLBCL.
* Adequate organ functions.
* Able to swallow capsules.

Exclusion Criteria:

* More than 3 prior treatments for this disease.
* Serious heart problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2002-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Royal Oak, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant Flow is reporting participants who discontinued from study drug. Per the protocol, a participant completed the study if the planned duration of treatment (6 cycles) was completed in the absence of disease progression or other reasons for discontinuation.
Groups:
- Enzastaurin: 500 milligrams (mg) enzastaurin (LY317615) tablets were administered in the morning within 30 minutes following a meal for 28 days (1 cycle) to be continued for up to 6 cycles in the absence of disease progression.
Period: Overall Study
Arm/Group | Enzastaurin
Started | 55
Received at Least 1 Dose of Study Drug | 55
Completed at Least 1 Cycle of Study Drug | 42
Completed | 1
Not Completed | 54
Not completed — Adverse Event | 2
Not completed — Death | 4
Not completed — Protocol Violation | 1
Not completed — Participant/Physician Perception | 1
Not completed — Progressive Disease | 41
Not completed — Other | 1
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Enzastaurin: 500 mg enzastaurin (LY317615) tablets were administered in the morning within 30 minutes following a meal for 28 days (1 cycle) to be continued for up to 6 cycles in the absence of disease progression.
Arm/Group | Enzastaurin
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50
  Black or African American | 2
  Asian | 1
  Hispanic | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55
PKCβ expression by IHC in DLBCL Tumors [Count of Participants; unit: Participants] — Protein Kinase C Beta (PKCβ) and Diffuse Large B-Cell Lymphoma (DLBCL). Protein expression was measured using an Immunohistochemistry (IHC) assay from tumor tissue samples that were scored using a 0 (negative, no staining) to 3+ (brightest staining) scoring system for cytoplasmic and nuclear staining. Three (3) participants had diagnostic tissue samples available for assay.
  Participants
    PKCβ Negative | 1
    PKCβ +1 | 1
    PKCβ +3 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Relapsed or Refractory DLBCL Who Are Progression-Free for at Least 2 Cycles (28-Day Cycles) After Receiving Enzastaurin (LY317615) (Clinical Response Rate)
Description: Clinical Response Rate in participants with DLBCL was calculated as (number of participants who were progression-free for at least two 28-day cycles [clinical responder]) divided by (total number of participants analyzed) multiplied by 100. Progression free survival (PFS) defined as the time from randomization to the first observation of disease progression or death due to any cause. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v 1.0) as 20% increase in the sum of the of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Randomization to measured progressive disease (PD) up to 34.3 months
Population: All randomized participants who remained on study for at least 1 cycle of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 42
percentage of participants | 21.8 [11.8 to 35.0]

2. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Overall Response Rate)
Description: Overall response rate was defined as best study response (CR or PR) using modified Southwest Oncology Group (SWOG) Response criteria. CR defined as the disappearance of detectable clinical and radiographic evidence of disease; regression of lymph nodes, nodal masses and spleen to normal size and absence of lymphoma in bone marrow infiltrate. PR was defined as a ≥50% decrease in the sum of the products of their diameters (SPD) in the 6 largest dominant nodes or nodal masses; no increase in size in the other nodes or liver or spleen; regression of nodes/lesions in organs by ≥50% in the SPD; or no new disease sites. The percentage participants was calculated as: (number of participants with CR or PR) divided by (number of participants qualified for tumor response analysis) multiplied by 100.
Time Frame: Randomization to measured PD or death up to 34.3 months
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 55
percentage of participants | 3.64

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first observation of disease progression or death due to any cause. For participants not known to have died as of the data cut-off date and who did not have PD, PFS was censored at the date of last follow-up visit. Progression is determined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v 1.0) as 20% increase in the sum of the of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Randomization to PD or death due to any cause up to 34.3 months
Population: All randomized participants who received at least 1 dose of study drug. Five (5) participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin
Number analyzed (Participants) | 55
months | 1.51 [1.02 to 1.74]

4. Secondary Outcome: Duration of Overall Response (DOR)
Description: Duration of CR or PR was defined as the time from first objective assessment to first time of disease progression or death from any cause using the modified SWOG Response criteria. CR defined as the disappearance of detectable clinical and radiographic evidence of disease, regression of lymph nodes, nodal masses and spleen to normal size and absence of lymphoma in bone marrow infiltrate. PR was defined as a ≥50% decrease in the SPD in the 6 largest dominant nodes or nodal masses, no increase in size in the other nodes, liver or spleen, regression of nodes/lesions in organs by ≥50% in the SPD, and no new disease sites. PD defined as >50% increase in SPD of the dominant nodal/non-nodal sites or new lesions. For participants who died, the duration of response was censored at death. For participants still alive, duration of overall response was censored at the last visit or follow-up visit. DOR was not analyzed due to low number of responders (CR or PR).
Time Frame: Time of response to PD up to 34.3 months
Population: Zero participants were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin
Number analyzed (Participants) | 2
months | NA [NA to NA] — Insufficient number of participants with events

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) or Who Died
Description: Clinically significant events were defined as serious AEs (SAEs) and other non-serious AEs. Participants who died due to PD, AEs while on treatment or died during the 30-day post-treatment period are included. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Randomization to study completion [Baseline up to 37 cycles (28-day cycles, 34.3 months) and 30-day follow-up]
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Enzastaurin: 500 mg enzastaurin (LY317615) was administered orally at dose in the morning within 30 minutes following a meal for 28 days (1 cycle) to be continued for up to 6 cycles in the absence of disease progression.
Arm/Group | Enzastaurin
Number analyzed (Participants) | 55
Participants
  Non-serious AEs | 51
  Serious AEs | 21
  Deaths Due to PD | 3
  Deaths Due to AEs | 1
  Deaths in 30-day follow-up | 11

6. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve at Steady State for One Dosing Interval (AUC0-24,ss) of Enzastaurin and Its Metabolite LY326020
Description: AUC0-24,ss during 1 dosing interval at steady state for Enzastaurin and its metabolite LY326020.
Time Frame: Cycle 1 Day 1 predose, 1 to 4 hours postdose and Cycle 1 Day 28 predose and at least 1-hour postdose (28-day cycle)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data to calculate AUC0-24,ss.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles*hour per liter (nmol*h/L)
Arm/Group | Enzastaurin
Number analyzed (Participants) | 33
nanomoles*hour per liter (nmol*h/L)
  Enzastaurin | 14800 (83.2)
  LY326020 | 14200 (39.6)

7. Secondary Outcome: PKCβ Expression by IHC in Readily Assessable DLBCL Tumors From Participants
Description: Protein expression was measured (cytoplasmic staining) using an IHC assay from a small subset of tumor tissue samples that were scored using a 0 (negative, no staining) to 3+ (brightest staining) scoring system, where higher staining indicated a greater PKCβ expression.
Time Frame: Baseline
Population: Participants who had paired diagnositic and relapsed tumor assessed for PKCβ expression.
Measure: Number; unit: participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 3
participants
  2+ at Diagnosis and 2+ at Relapse | 1
  0 at Diagnosis and 1+ at Relapse | 1
  3+ and 0 at Diagnosis and 3+ at Relapse | 1

ADVERSE EVENTS:
Description: Study-specific clinical outcomes due to PD were not considered to be a SAE unless the investigator deemed it related to the use of the study drug.
Groups:
- Enzastaurin: 500 mg enzastaurin tablets were administered in the morning within 30 minutes of a meal for 28 days (1 cycle) to be continued for up to 6 cycles in the absence of disease progression.
Arm/Group | Enzastaurin
Serious Adverse Events (participants affected / at risk) | 21/55
Other Adverse Events (participants affected / at risk) | 51/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=55)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Clostridium difficile sepsis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2)
Azotaemia (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=55)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 10 (12)
Flatulence (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 15 (15)
Vomiting (Gastrointestinal disorders) | 11 (11)
Asthenia (General disorders) | 5 (5)
Chills (General disorders) | 5 (5)
Fatigue (General disorders) | 18 (21)
Oedema (General disorders) | 5 (5)
Oedema peripheral (General disorders) | 13 (16)
Pyrexia (General disorders) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 4 (7)
Urinary tract infection (Infections and infestations) | 3 (3)
Blood creatinine increased (Investigations) | 4 (4)
Weight decreased (Investigations) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Dizziness (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4)
Chromaturia (Renal and urinary disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Night sweats (Skin and subcutaneous tissue disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days